CLINICAL TRIAL: NCT00063570
Title: Phase II Trial of Alimta (Pemetrexed) and Gemzar (Gemcitabine) in Metastatic Breast Cancer Patients Who Have Received Prior Taxane Therapy
Brief Title: Pemetrexed Plus Gemcitabine in Metastatic Breast Cancer Patients After Receiving Taxane Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5141; H3E-US-JMEO
Record Dates: First submitted 2003-06-30; First posted 2003-07-01 (Estimated); Results first posted 2009-05-13 (Estimated); Last update posted 2009-05-29 (Estimated); Status verified 2009-05

CONDITIONS: Breast Cancer; Breast Neoplasms
Keywords: Cancer of Breast; Cancer of the Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — Pemetrexed; Gemcitabine

ARMS (2):
- A (Experimental)
  Interventions: Drug: Pemetrexed; Drug: Gemcitabine
- B (Experimental)
  Interventions: Drug: Gemcitabine; Drug: Pemetrexed

INTERVENTIONS:
Drug: Pemetrexed — 500 mg/m2, intravenous (IV), every 14 days, until disease progression
  Other Names: LY231514, Alimta
  Arms: A
Drug: Gemcitabine — 1500 mg/m2, intravenous (IV), every 14 days, until disease progression
  Other Names: LY188011, Gemzar
  Arms: A
Drug: Gemcitabine — 1000 mg/m2, intravenous (IV), on Days 1 and 8 of 21-day cycle, until disease progression
  Other Names: LY188011; Gemzar
  Arms: B
Drug: Pemetrexed — 500 mg/m2, intravenous (IV), every 21 days, until disease progression
  Other Names: LY231514; Alimta
  Arms: B

SUMMARY:
The purpose of the study is to determine if the two drugs can help patients feel better while causing the tumor to become smaller or disappear; evaluate the safety of giving both pemetrexed and gemcitabine in patients with advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Must have received prior chemotherapy with Taxol (paclitaxel) or Taxotere (docetaxel).
* Less than 3 different chemotherapy treatments for metastatic disease.
* Prior treatment with hormonal and/or radiation therapy.
* Must have disease that can be measured.
* Must be able to take care of self needs for example personal hygiene

Exclusion Criteria:

* Must not be pregnant or breast-feeding.
* Cancer that has spread to the brain.
* Treatment with Gemcitabine or Pemetrexed
* Unable to take folic acid or Vitamin B12
* Treatment for another cancer within the last 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2003-07; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 317-615-4559 Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- United States (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Aurora, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Plantation, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Morrisville, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Seattle, Washington
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician., San Juan, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: At completion of the first stage of the trial, toxicities associated with the Day 8 dosing of gemcitabine were observed, and the protocol was amended to a bi-weekly schedule. Patients were analyzed separately according to the study drug schedule received.
Groups:
- Bi-Weekly Schedule: Pemetrexed: 500 mg/m2, intravenous (IV), every 14 days, until disease progression.
  Gemcitabine: 1500 mg/m2, intravenous (IV), every 14 days, until disease progression.
- 21-Day Schedule: Pemetrexed: 500 mg/m2, intravenous (IV), every 21 days, until disease progression.
  Gemcitabine: 1000 mg/m2, intravenous (IV) on Days 1 and 8 of a 21-day cycle, until disease progression.
Period: Overall Study
Arm/Group | Bi-Weekly Schedule | 21-Day Schedule
Started | 52 | 21
Completed | 52 (Completed for this study means patient received study drug and was eligible for efficacy analysis.) | 21 (Completed for this study means patient received study drug and was eligible for efficacy analysis.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bi-Weekly Schedule | 21-Day Schedule | Total
Number analyzed (Participants) | 52 | 21 | 73
Age Continuous [Median (Full Range); unit: years] | 53.5 [33 to 73] | 50.7 [28 to 73] | 51.9 [28 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 21 | 73
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 52 | 21 | 73
Current Pathological Diagnosis [Number; unit: paticipants]
  Ductal breast carcinoma | 36 | 12 | 48
  Lobular breast carcinoma | 2 | 0 | 2
  Adenocystic breast carcinoma | 0 | 1 | 1
  Breast carcinoma | 4 | 4 | 8
  Other | 7 | 3 | 10
  Unknown | 1 | 1 | 2
  No current pathological diagnosis | 2 | 0 | 2
Karnofsky Performance Status (KPS) [Number; unit: participants] — The Karnofsky Performance Status Index classifies functional impairment. Scores range from 0 to 100. A higher score means the patient is better able to carry out daily activities.
  participants
    <=60 - Needs increasing assistance up to Death (0) | 0 | 0 | 0
    70 - Unable to carry on normal activity | 4 | 1 | 5
    80 - Activity with effort; some signs of disease | 11 | 5 | 16
    90 - Normal activity; minor signs of disease | 19 | 9 | 28
    100 - Normal no complaints; no evidence of disease | 17 | 6 | 23
    unknown | 1 | 0 | 1
Menopausal Status at Cycle 0 [Number; unit: participants]
  Pre-Menopausal | 7 | 3 | 10
  Menopausal | 4 | 3 | 7
  Post-Menopausal | 41 | 15 | 56
Patients with Current Pathological Diagnosis [Number; unit: participants]
  Yes | 50 | 21 | 71
  No | 2 | 0 | 2
Race/Ethnicity [Number; unit: participants]
  Caucasian | 44 | 20 | 64
  African | 4 | 1 | 5
  East/Southeast Asian | 3 | 0 | 3
  Hispanic | 1 | 0 | 1
Time (in months) from Current Pathological Diagnosis to Enrollment [Median (Full Range); unit: Months] | 13.08 [0.4 to 134.2] | 14.31 [0.5 to 57.1] | 14.29 [0.4 to 134.2]

OUTCOME MEASURES:

1. Primary Outcome: Overall Tumor Response
Description: Best overall (confirmed) response recorded from start of treatment until disease progression/recurrence, start of other anti-tumor therapy/intervention, or end of trial, whichever comes first. Response must be confirmed at least 6 weeks from previous scans. Best overall response assignment depends on both measurement and confirmation criteria.
Time Frame: Every 6 weeks from start of treatment until documented disease progression or for 6 months from last dose of study drug, whichever occurs first. After 6 months, clinical assessment every 12 weeks and radiologic test performed as clinically indicated
Population: Patients who received at least one dose of study drug (pemetrexed or gemcitabine) were included in the analyses.
Measure: Number; unit: participants
Arm/Group | Bi-Weekly Schedule | 21-Day Schedule
Number analyzed (Participants) | 52 | 21
participants
  Complete Response | 2 | 0
  Partial Response | 8 | 5
  Stable Disease | 26 | 10
  Progressive Disease | 14 | 6
  Unknown | 2 | 0

2. Secondary Outcome: Duration of (Confirmed) Complete Response or Partial Response
Description: Duration of response is calculated as (Date of First Disease Progression or Death as a Result of any Cause whichever Comes First - Date of First Objective Status Assessment of Confirmed CR or PR + 1)/(365.25/12).
Time Frame: as for outcome 1
Population: Number of patients with a confirmed complete or partial response.
Measure: Median (Full Range); unit: months
Arm/Group | Bi-Weekly Schedule | 21-Day Schedule
Number analyzed (Participants) | 10 | 5
months | 5.85 [2.79 to 16.79] | 4.17 [3.71 to 17.61]

3. Secondary Outcome: Time to Progressive Disease
Description: Time to progressive disease is calculated as (Date of First Disease Progression or Death Due to Disease under Study whichever Comes First - First Dose Date + 1)/(365.25/12).
Time Frame: as for outcome 1
Population: Intention to Treat analysis
Measure: Median (Full Range); unit: months
Arm/Group | Bi-Weekly Schedule | 21-Day Schedule
Number analyzed (Participants) | 52 | 21
months | 3.19 [0.16 to 18.20] | 4.01 [1.05 to 20.80]

4. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure is calculated as (Date of First Disease Progression, Death as a Result of any Cause, or Early Discontinuation of Treatment Due to Adverse Event or Physician Perception of Lack of Efficacy or Patient and Physician Perception of Lack of Efficacy, whichever Comes First - First Dose Date + 1)/ (365.25/12)
Time Frame: as for outcome 1
Population: Intention to Treat analysis
Measure: Median (Full Range); unit: months
Arm/Group | Bi-Weekly Schedule | 21-Day Schedule
Number analyzed (Participants) | 52 | 21
months | 2.79 [0.16 to 18.20] | 2.56 [0.49 to 20.80]

5. Secondary Outcome: Overall Survival
Description: Overall survival time is calculated as (Date of Death as a Result of any Cause - First Dose Date + 1)/ (365.25/12).
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: months
Arm/Group | Bi-Weekly Schedule | 21-Day Schedule
Number analyzed (Participants) | 52 | 21
months | 13.44 [0.76 to 36.60] | 16.20 [1.41 to 31.64]

ADVERSE EVENTS:
Arm/Group | Bi-Weekly Schedule | 21-Day Schedule
Serious Adverse Events (participants affected / at risk) | 17 | 7
Other Adverse Events (participants affected / at risk) | 51 | 21
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Bi-Weekly Schedule | 21-Day Schedule
Anaemia (Blood and lymphatic system disorders) | 2/52 (2) | 0/21 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 4/52 (5) | 1/21 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1/52 (1) | 0/21 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0/52 (0) | 1/21 (1)
Abdominal pain (Gastrointestinal disorders) | 1/52 (1) | 0/21 (0)
Constipation (Gastrointestinal disorders) | 1/52 (1) | 0/21 (0)
Pyrexia (General disorders) | 2/52 (3) | 1/21 (1)
Hepatic failure (Hepatobiliary disorders) | 1/52 (2) | 0/21 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1/52 (1) | 0/21 (0)
Device related infection (Infections and infestations) | 1/52 (1) | 0/21 (0)
Pneumonia (Infections and infestations) | 2/52 (2) | 0/21 (0)
Sepsis (Infections and infestations) | 1/52 (1) | 0/21 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0/52 (0) | 1/21 (1)
Fracture (Injury, poisoning and procedural complications) | 1/52 (1) | 0/21 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1/52 (1) | 0/21 (0)
Drug level increased (Investigations) | 1/52 (1) | 0/21 (0)
Dehydration (Metabolism and nutrition disorders) | 2/52 (2) | 0/21 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1/52 (1) | 0/21 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 1/52 (1) | 0/21 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/52 (1) | 0/21 (0)
Convulsion (Nervous system disorders) | 1/52 (1) | 0/21 (0)
Dizziness (Nervous system disorders) | 0/52 (0) | 1/21 (1)
Lumbar radiculopathy (Nervous system disorders) | 1/52 (1) | 0/21 (0)
Meningitis noninfective (Nervous system disorders) | 1/52 (1) | 0/21 (0)
Mental status changes (Psychiatric disorders) | 1/52 (1) | 0/21 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0/52 (0) | 1/21 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1/52 (1) | 0/21 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2/52 (2) | 0/21 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1/52 (1) | 0/21 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0/52 (0) | 1/21 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0/52 (0) | 1/21 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1/52 (1) | 0/21 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1/52 (1) | 0/21 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0/52 (0) | 1/21 (1)
Aortic stenosis (Vascular disorders) | 0/52 (0) | 1/21 (1)
Superior vena caval occlusion (Vascular disorders) | 0/52 (0) | 1/21 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Bi-Weekly Schedule | 21-Day Schedule
Anaemia (Blood and lymphatic system disorders) | 23/52 (40) | 12/21 (22)
Febrile neutropenia (Blood and lymphatic system disorders) | 2/52 (2) | 3/21 (3)
Leukopenia (Blood and lymphatic system disorders) | 13/52 (18) | 6/21 (22)
Lymphopenia (Blood and lymphatic system disorders) | 1/52 (2) | 2/21 (10)
Neutropenia (Blood and lymphatic system disorders) | 23/52 (35) | 16/21 (53)
Thrombocythaemia (Blood and lymphatic system disorders) | 1/52 (1) | 2/21 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 10/52 (14) | 8/21 (20)
Tachycardia (Cardiac disorders) | 5/52 (5) | 1/21 (1)
Diplopia (Eye disorders) | 0/52 (0) | 2/21 (4)
Eye irritation (Eye disorders) | 4/52 (4) | 3/21 (4)
Eye swelling (Eye disorders) | 3/52 (3) | 0/21 (0)
Lacrimation increased (Eye disorders) | 8/52 (9) | 1/21 (1)
Vision blurred (Eye disorders) | 3/52 (3) | 0/21 (0)
Abdominal discomfort (Gastrointestinal disorders) | 3/52 (3) | 0/21 (0)
Abdominal distension (Gastrointestinal disorders) | 5/52 (7) | 3/21 (3)
Abdominal pain (Gastrointestinal disorders) | 10/52 (13) | 5/21 (6)
Abdominal pain upper (Gastrointestinal disorders) | 5/52 (6) | 0/21 (0)
Constipation (Gastrointestinal disorders) | 26/52 (40) | 6/21 (11)
Diarrhoea (Gastrointestinal disorders) | 16/52 (18) | 12/21 (14)
Dry mouth (Gastrointestinal disorders) | 3/52 (6) | 0/21 (0)
Dyspepsia (Gastrointestinal disorders) | 5/52 (5) | 3/21 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6/52 (6) | 0/21 (0)
Haemorrhoids (Gastrointestinal disorders) | 3/52 (3) | 2/21 (2)
Nausea (Gastrointestinal disorders) | 28/52 (46) | 14/21 (28)
Stomatitis (Gastrointestinal disorders) | 9/52 (12) | 3/21 (4)
Vomiting (Gastrointestinal disorders) | 10/52 (13) | 7/21 (16)
Asthenia (General disorders) | 6/52 (9) | 4/21 (6)
Chest discomfort (General disorders) | 3/52 (5) | 1/21 (2)
Chest pain (General disorders) | 4/52 (4) | 4/21 (5)
Chills (General disorders) | 7/52 (9) | 6/21 (7)
Face oedema (General disorders) | 4/52 (4) | 0/21 (0)
Fatigue (General disorders) | 35/52 (68) | 15/21 (28)
Feeling hot (General disorders) | 0/52 (0) | 2/21 (2)
Mucosal inflammation (General disorders) | 6/52 (7) | 4/21 (4)
Oedema (General disorders) | 5/52 (6) | 1/21 (1)
Oedema peripheral (General disorders) | 12/52 (15) | 4/21 (5)
Pain (General disorders) | 5/52 (6) | 3/21 (4)
Pyrexia (General disorders) | 15/52 (23) | 14/21 (25)
Hypersensitivity (Immune system disorders) | 3/52 (4) | 0/21 (0)
Cellulitis (Infections and infestations) | 3/52 (3) | 0/21 (0)
Sinusitis (Infections and infestations) | 3/52 (3) | 2/21 (2)
Upper respiratory tract infection (Infections and infestations) | 5/52 (7) | 3/21 (3)
Urinary tract infection (Infections and infestations) | 4/52 (6) | 1/21 (1)
Alanine aminotransferase increased (Investigations) | 12/52 (15) | 7/21 (17)
Aspartate aminotransferase increased (Investigations) | 14/52 (17) | 9/21 (19)
Blood alkaline phosphatase increased (Investigations) | 6/52 (6) | 5/21 (7)
Haemoglobin decreased (Investigations) | 4/52 (5) | 2/21 (7)
Neutrophil count decreased (Investigations) | 2/52 (2) | 4/21 (4)
Weight decreased (Investigations) | 3/52 (3) | 0/21 (0)
White blood cell count decreased (Investigations) | 0/52 (0) | 3/21 (5)
Anorexia (Metabolism and nutrition disorders) | 10/52 (11) | 8/21 (12)
Decreased appetite (Metabolism and nutrition disorders) | 2/52 (3) | 2/21 (2)
Dehydration (Metabolism and nutrition disorders) | 1/52 (1) | 2/21 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 11/52 (16) | 2/21 (10)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1/52 (1) | 2/21 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 2/52 (2) | 2/21 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 6/52 (9) | 6/21 (9)
Hyponatraemia (Metabolism and nutrition disorders) | 4/52 (5) | 3/21 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9/52 (11) | 6/21 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 8/52 (8) | 5/21 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 3/52 (4) | 3/21 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0/52 (0) | 2/21 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6/52 (6) | 1/21 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3/52 (5) | 4/21 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 7/52 (14) | 5/21 (16)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4/52 (5) | 6/21 (7)
Dizziness (Nervous system disorders) | 3/52 (3) | 4/21 (5)
Dysgeusia (Nervous system disorders) | 5/52 (8) | 2/21 (2)
Headache (Nervous system disorders) | 11/52 (17) | 11/21 (12)
Hypoaesthesia (Nervous system disorders) | 3/52 (3) | 3/21 (3)
Lethargy (Nervous system disorders) | 2/52 (2) | 2/21 (3)
Neuropathy peripheral (Nervous system disorders) | 3/52 (3) | 3/21 (3)
Paraesthesia (Nervous system disorders) | 3/52 (3) | 3/21 (4)
Sinus headache (Nervous system disorders) | 0/52 (0) | 2/21 (2)
Somnolence (Nervous system disorders) | 0/52 (0) | 2/21 (2)
Tremor (Nervous system disorders) | 3/52 (3) | 0/21 (0)
Anxiety (Psychiatric disorders) | 6/52 (6) | 3/21 (4)
Confusional state (Psychiatric disorders) | 4/52 (5) | 0/21 (0)
Insomnia (Psychiatric disorders) | 9/52 (9) | 3/21 (3)
Dysuria (Renal and urinary disorders) | 3/52 (3) | 1/21 (1)
Breast pain (Reproductive system and breast disorders) | 1/52 (1) | 2/21 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 14/52 (15) | 7/21 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15/52 (20) | 6/21 (10)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5/52 (6) | 0/21 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5/52 (5) | 2/21 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3/52 (3) | 0/21 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3/52 (3) | 0/21 (0)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 3/52 (5) | 4/21 (4)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2/52 (2) | 5/21 (9)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2/52 (2) | 2/21 (3)
Acne (Skin and subcutaneous tissue disorders) | 0/52 (0) | 2/21 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 8/52 (8) | 3/21 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 5/52 (6) | 1/21 (1)
Erythema (Skin and subcutaneous tissue disorders) | 5/52 (6) | 4/21 (9)
Night sweats (Skin and subcutaneous tissue disorders) | 5/52 (5) | 3/21 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 9/52 (10) | 4/21 (6)
Rash (Skin and subcutaneous tissue disorders) | 23/52 (30) | 15/21 (18)
Rash macular (Skin and subcutaneous tissue disorders) | 3/52 (4) | 1/21 (1)
Flushing (Vascular disorders) | 1/52 (1) | 6/21 (6)
Lymphoedema (Vascular disorders) | 6/52 (9) | 2/21 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days